CLINICAL TRIAL: NCT04725890
Title: Safety and Feasibility of Endoscopic Application of a Novel Therapy for Duodenal Mucosal Regeneration in the Treatment of Type II Diabetes
Brief Title: Safety and Feasibility of a Novel Endoscopic Intervention for the Treatment of Type II Diabetes
Acronym: REGENT-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endogenex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 196
Record Dates: First submitted 2021-01-18; First posted 2021-01-27 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Intervention (Experimental): All eligible participants will receive the DyaMX procedure.
  Interventions: Device: The DyaMX Device

INTERVENTIONS:
Device: The DyaMX Device — The DyaMX device is designed to induce duodenal mucosal regeneration using pulsed electric field. The DyaMX procedure is a non-surgical, endoscopic procedure.
  Other Names: Duodenal Mucosal Regeneration

SUMMARY:
This is an open-label study to assess the safety and feasibility of the DyaMX device for endoscopic duodenal mucosal regeneration in individuals with type 2 diabetes inadequately controlled on glucose-lowering medications.

DETAILED DESCRIPTION:
Individuals who sign the informed consent will be screened for study eligibility. Eligible participants will be treated with the DyaMX procedure and followed up for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years of age
2. Current diagnosis of T2D
3. History of T2D for less than or equal to 10 years, or use insulin for less or equal to 10 years
4. HbA1C of 7.5-11.0%
5. BMI 24-40 kg/m2
6. If treated with non-insulin glucose lowering mediations, the medications (1-4 medications) should be stable for at least 12 weeks prior to baseline visit. If treated with basal insulin, the daily insulin dose should be within 20-60 IU.
7. Agree not to donate blood during participation in the study.
8. If treated with non-insulin glucose lowering medications, participant should have weight stability (defined as a < 5% change in body weight) for at least 12 weeks prior to the screening visit
9. Able to comply with study requirements and understand and sign the Informed Consent Form
10. Women of childbearing potential must be using an acceptable method of contraception throughout the study
11. Willing and able to perform self-monitoring blood glucose and comply with study visits and study tasks as required per protocol.

Exclusion Criteria:

1. Diagnosed with type 1 diabetes
2. History of diabetic ketoacidosis or hyperosmolar nonketotic coma
3. Probable insulin production failure, defined as overnight fasting C-peptide serum <1 ng/mL (333pmol/l).
4. Previous use of any types of insulin for >1 month (at any time, except for treatment of gestational diabetes) in last 2 years for those on non-insulin medications.
5. Current use of multiple daily dose insulin or insulin pump
6. Hypoglycemia unawareness
7. History of ≥1 severe hypoglycemia (defined by needing for third-party assistance), unless a clear correctable precipitating factor can be identified, in past 6 months from the screening visit
8. Known autoimmune disease, as evidenced by a positive anti-glutamic acid decarboxylase (GAD) test, including but not limited to celiac disease, or pre-existing symptoms of systemic lupus erythematosus, scleroderma or other autoimmune connective tissue disorder.
9. Previous GI surgery that has changed GI anatomy or could limit treatment of the duodenum, such as Billroth 2, Roux-en-Y gastric bypass, gastric band or other similar procedures or conditions.
10. Known history of a structural or functional disorder of the upper GI tract that may impede passage of the device through the upper GI tract or increase risk of tissue damage during an endoscopic procedure, including esophagitis, stricture/stenosis, varices, diverticula, or other disorder of the esophagus, stomach and duodenum.
11. Active H. pylori infection (Participants with active H. pylori may continue with the screening process if they are treated with an appropriate antibiotic regimen)
12. History of, or gastrointestinal symptoms suggestive of gastroparesis.
13. Acute gastrointestinal illness in the previous 7 days
14. Known history irritable bowel syndrome, radiation enteritis or other inflammatory bowel disease, such as Crohn's disease and Celiac disease
15. History of chronic or acute pancreatitis.
16. Known active hepatitis or active liver disease other than NASH/NAFLD.
17. Alcoholic liver disease, as indicated by ANI >0
18. Current use of anticoagulation therapy (such as warfarin) that cannot be discontinued for 7 days before and 14 days after the procedure.
19. Current use of P2Y12 inhibitors (clopidogrel, prasugrel, ticagrelor) that cannot be discontinued for 14 days before and 14 days after the procedure.
20. Unable to discontinue non-steroidal anti-inflammatory drugs (NSAIDs) during treatment through 4 weeks following the procedure. Use of acetaminophen and low dose aspirin is allowed.
21. Use of systemic glucocorticoids (excluding topical or ophthalmic application or inhaled forms) for more than 10 consecutive days within 12 weeks prior to the baseline visit.
22. Use of drugs known to affect GI motility (e.g. Metoclopramide)
23. Use of weight loss medications such as Phentermine, Meridia, Xenical, or over-the-counter weight loss medications (prescription medication)
24. Persistent anemia, defined as hemoglobin <10 g/dL.
25. Known history of blood donation or transfusion within 3 months prior to the Screening Visit.
26. Known history of cardiac arrhythmia
27. Significant cardiovascular disease, including known history of valvular disease, or myocardial infarction, heart failure, transient ischemic attack, or stroke within 6 months prior to the Screening Visit.
28. Estimated glomerular filtration rate (eGFR) ≤ 30 ml/min/1.73m2.
29. Known immunocompromised status, including but not limited to individuals who have undergone organ transplantation, chemotherapy, or radiotherapy within the past 12 months, who have clinically-significant leukopenia, who are positive for the human immunodeficiency virus (HIV) or whose immune status makes the participant a poor candidate for clinical trial participation in the opinion of the investigator.
30. With any implanted electronic devices or duodenal metallic implants
31. Not a candidate for upper GI endoscopy or general anesthesia.
32. Active illicit substance abuse or alcoholism (> 2 drinks/day regularly).
33. Active malignancy within the last 5 years (excluding non-melanoma skin cancers)
34. Women breast feeding
35. Participating in another ongoing clinical trial of an investigational drug or device.
36. Any other mental or physical condition which, in the opinion of the study investigator, makes the participant a poor candidate for clinical trial participation.
37. Critically ill or has a life expectancy <3 years

    Additional exclusion criteria to be confirmed during the screening process:
38. HbA1c < 7.5% or > 11% at baseline visit
39. Any severe hypoglycemic event since the screening visit
40. Glucose level <54 mg/dl (3.0 mmol/l) in more than 1% of time by CGM since the screening visit
41. Uncontrolled hyperglycemia with a glucose level >270 mg/dl (>15 mmol/L) after an overnight fast or >360 mg/dl (>20 mmol/l) in a randomly performed measurement that is confirmed by a second measurement (not on the same day) since screening visit
42. Mean of 3 separate blood pressure measurements >180 mmHg (systolic) or >100 mmHg (diastolic)
43. Women of child-bearing potential with a positive urine pregnancy test at baseline visit
44. Grade III or greater esophagitis on endoscopy
45. Abnormalities of the GI tract preventing endoscopic access to the duodenum
46. Anatomic abnormalities in the duodenum that would preclude the completion of the treatment procedure, including tortuous anatomy
47. Endoscopic observation of upper gastrointestinal abnormality such as ulcers, polyps, varices, strictures, congenital or intestinal telangiectasia
48. Any other anatomical or endoscopic abnormalities/characteristics that, in the opinion of the investigator, would preclude safe use of the investigational device or procedure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Sartoretto, MD, Principal Investigator — The BMI Clinic
Locations (2):
- Australia (2):
  - The BMI Clinic, Sydney, New South Wales
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 3 medical centers in Australia between January of 2021 and November of 2023. Participants were considered enrolled in the study once they passed endoscopic screening. Screen failures were defined as participants who consented for the study, started the screening process but were not subsequently enrolled. The first participant was enrolled on 20-Apr-2021 and the last on 27-Jul-2023.
Pre-assignment Details: A total of 65 participants were enrolled in the study.
Groups:
- Intervention- Endogenex (PEF) Treatment: Enrolled participants include all eligible participants that met inclusion criteria and did not meet any exclusion criteria and were treated with the Endogenex/DyaMX device. The Endogenex/DyaMX device is designed to induce duodenal mucosal regeneration using pulsed electric field via a non-surgical, endoscopic procedure.
Period: Overall Study
Arm/Group | Intervention- Endogenex (PEF) Treatment
Started | 65
Completed | 59
Not Completed | 6
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Intervention- Non-Insulin Cohort: Non-insulin Arm: All participants are on at least one non-insulin, glucose-lowering medications and received the Endogenex treatment
- Intervention- Insulin Cohort: Insulin (IS) Cohort: all participants are on insulin and received the Endogenex treatment.
- Total: Total of all reporting groups
Arm/Group | Intervention- Non-Insulin Cohort | Intervention- Insulin Cohort | Total
Number analyzed (Participants) | 51 | 14 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (8.0) | 58.1 (7.0) | 53.9 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 21
  Male | 38 | 6 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 49 | 14 | 63
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 2 | 13
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 1 | 1
  White | 35 | 6 | 41
  More than one race | 4 | 5 | 9
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 51 | 14 | 65
HbA1c [Mean (Standard Deviation); unit: %] — The unit of measure for HbA1c is %.
  % | 8.8 (0.9) | 8.5 (0.8) | 8.7 (0.9)
Weight [Mean (Standard Deviation); unit: Kg] | 93.6 (15.4) | 80.2 (11.8) | 90.7 (15.6)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 31.5 (3.5) | 29.5 (4.2) | 31.1 (3.7)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 10.1 (2.7) | 8.6 (1.6) | 9.7 (2.3)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 5.5 (2.4) | 12.4 (5.4) | 7.0 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Device- or Procedure-related Serious Adverse Events (SAE)
Description: Number of participants experiencing one or more device- or procedure-related serious adverse events at 12 weeks post procedure
Time Frame: At 12 weeks post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention- Non-Insulin Cohort | Intervention- Insulin Cohort
Number analyzed (Participants) | 51 | 14
Participants | 0 | 1

2. Secondary Outcome: HbA1c by Post Procedure Follow-up Visit
Description: Mean HbA1c (%) by Post Procedure Follow-up Visit. The unit of measure for HbA1c is %.
Time Frame: Follow up at 12, 24, and 48 weeks post procedure
Population: The unit of measure for HbA1c is %. Six participants were exited from the study. For the IS Cohort, one of the 6 was exited prior to 12 weeks and one participant missed the 24 week visit. In the NIS Cohort, two were exited prior to the 24 week visit and three after the 24 week visit/prior to the 48 week visit. Two additional NIS participants missed their 24 week visit.
Measure: Mean (Standard Deviation); unit: HbA1c %
Arm/Group | Intervention- Non-Insulin Cohort | Intervention- Insulin Cohort
Number analyzed (Participants) | 51 | 14
HbA1c %
  Mean HbA1c at Baseline | 8.8 (0.9) | 8.5 (0.8)
  Mean HbA1c at 12 Weeks: number analyzed (Participants) | 51 | 13
  Mean HbA1c at 12 Weeks | 7.7 (1.2) | 7.9 (0.99)
  Mean HbA1c at 24 Weeks: number analyzed (Participants) | 47 | 12
  Mean HbA1c at 24 Weeks | 7.8 (2.4) | 8.1 (1.0)
  Mean HbA1c at 48 Weeks: number analyzed (Participants) | 46 | 13
  Mean HbA1c at 48 Weeks | 7.7 (2.4) | 7.6 (1.0)

3. Secondary Outcome: Fasting Plasma Glucose by Visit
Description: Mean Fasting Plasma Glucose by Visit
Time Frame: Baseline, 12, 24, and 48 weeks
Population: Six participants were exited from the study. For the IS Cohort, one of the 6 was exited prior to 12 weeks and one participant missed the 24 week visit. In the NIS Cohort, two were exited prior to the 24 week visit and three after the 24 week visit/prior to the 48 week visit. Two additional participants missed their 24 week visit.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Intervention- Non-Insulin Cohort | Intervention- Insulin Cohort
Number analyzed (Participants) | 51 | 14
mmol/L
  Mean FPG at Baseline | 10.1 (2.7) | 8.6 (1.6)
  Mean FPG at 12 Weeks: number analyzed (Participants) | 51 | 13
  Mean FPG at 12 Weeks | 8.4 (2.3) | 8.3 (2.3)
  Mean FPG at 24 Weeks: number analyzed (Participants) | 47 | 12
  Mean FPG at 24 Weeks | 7.6 (2.6) | 8.8 (2.9)
  Mean FPG at 48 Weeks: number analyzed (Participants) | 46 | 13
  Mean FPG at 48 Weeks | 7.9 (3.1) | 7.5 (1.9)

4. Secondary Outcome: Weight by Visit
Description: Mean Weight by Visit
Time Frame: Baseline, 12, 24, and 48 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Intervention- Non-Insulin Cohort | Intervention- Insulin Cohort
Number analyzed (Participants) | 51 | 14
kg
  Mean Weight at Baseline | 94 (15) | 80 (12)
  Mean Weight at 12 Weeks: number analyzed (Participants) | 51 | 13
  Mean Weight at 12 Weeks | 90 (14) | 79 (11)
  Mean Weight at 24 Weeks: number analyzed (Participants) | 47 | 12
  Mean Weight at 24 Weeks | 86 (32) | 77 (12)
  Mean Weight at 48 Weeks: number analyzed (Participants) | 46 | 13
  Mean Weight at 48 Weeks | 89 (30) | 73 (12)

5. Other Pre Specified Outcome: Procedural Success
Description: Percentage of participants with successful DMR procedure
Time Frame: At the time of the Index Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention- Non-Insulin Cohort | Intervention- Insulin Cohort
Number analyzed (Participants) | 51 | 14
Participants | 51 | 14

6. Other Pre Specified Outcome: Procedural Time
Description: Time between catheter insertion to catheter removal
Time Frame: Time of Procedure
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Intervention- Non-Insulin Cohort | Intervention- Insulin Cohort
Number analyzed (Participants) | 51 | 14
Minutes | 74.3 (31.7) | 102.5 (36.5)

ADVERSE EVENTS:
Time Frame: Baseline through 48 Weeks (duration of the study)
Arm/Group | Intervention- Endogenex (PEF) Treatment
All-Cause Mortality (participants affected / at risk) | 0/65
Serious Adverse Events (participants affected / at risk) | 5/65
Other Adverse Events (participants affected / at risk) | 58/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention- Endogenex (PEF) Treatment (N=65)
Colon Cancer (Gastrointestinal disorders) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Celiac Artery stenosis (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention- Endogenex (PEF) Treatment (N=65)
COVID-19 (Infections and infestations) | 26 (26)
Oropharyngeal pain (Gastrointestinal disorders) | 26 (26)
Diarrhea (Gastrointestinal disorders) | 15 (16)
Nausea (Gastrointestinal disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 6 (6)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5 (5)
Adverse Drug Reaction (General disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Flatulence (Gastrointestinal disorders) | 3 (3)
Headache (Nervous system disorders) | 3 (3)
Joint injury (Musculoskeletal and connective tissue disorders) | 3 (3)
Lip Injury (Injury, poisoning and procedural complications) | 3 (3)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 3 (3)
Respiratory tract infection (Infections and infestations) | 3 (3)
Upper respiratory tract infectio (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Candida infection (Infections and infestations) | 2 (2)
Cellulitis (Infections and infestations) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Gastrointestinal procedural complication (Injury, poisoning and procedural complications) | 2 (2)
Hyperglycemia (Endocrine disorders) | 2 (2)
Influenza (Infections and infestations) | 2 (2)
Injection site pain (General disorders) | 2 (2)
Lethargy (Gastrointestinal disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pyrexia (General disorders) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Vaccination complication (Immune system disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Anesthesia eye (Eye disorders) | 1 (1)
Back injury (Musculoskeletal and connective tissue disorders) | 1 (1)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dental caries (General disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Dizziness postural (Cardiac disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Hemorrhoidal hemorrhage (Vascular disorders) | 1 (1)
Helicobacter gastritis (Gastrointestinal disorders) | 1 (1)
Hepatic enzyme increased (Hepatobiliary disorders) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1)
Ketosis (Metabolism and nutrition disorders) | 1 (1)
Lactose intolerance (Metabolism and nutrition disorders) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Parainfluenza virus infection (Infections and infestations) | 1 (1)
Presyncope (Cardiac disorders) | 1 (1)
Pyelonephritis (Renal and urinary disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Infection (Skin and subcutaneous tissue disorders) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection bacterial (Infections and infestations) | 1 (1)
Urinary tract infection viral (Renal and urinary disorders) | 1 (1)
Viral Infection (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This pilot study was performed to provide an early assessment of safety of the Endogenex device in participants with Type 2 Diabetes. Due to the small sample size, formal hypothesis testing was not performed and data may be limited to descriptive statistics, including mean and standard deviations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-09-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT04725890/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT04725890/SAP_002.pdf